CLINICAL TRIAL: NCT04431258
Title: A Phase I Open Label Followed by a Phase II Randomized, Controlled Study to Assess the Efficacy and Safety of ABTL0812 in Combination With FOLFIRINOX for First-line Treatment of Metastatic Pancreatic
Brief Title: ABTL0812 in Combination With FOLFIRINOX for First-line Treatment of Metastatic Pancreatic Study
Acronym: PanC-ASAP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ability Pharmaceuticals SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ABT-C11-2020; 2020-002791-13 (EudraCT Number); FD-R-006817-01 (Other Grant/Funding Number: FDA OOPD)
Record Dates: First submitted 2020-05-27; First posted 2020-06-16 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — ABTL0812; folfirinox; Drug Therapy

STUDY DESIGN:
Intervention Model Description: Double blind, randomized, placebo-controlled, multicenter study
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A) ABTL0812 + FOLFIRINOX (Experimental): FOLFIRINOX will be dosed according to the standard following regimen:
  * oxaliplatin 85 mg/m2, administered as 2-hour iv infusion
  * leucovorin 400 mg/m2, administered as 2-hour iv infusion
  * irinotecan 180 mg/m2, administered as 1.5-hour iv infusion
  * fluorouracil 2400 mg/m2, administered as 46-hour iv infusion every 2 weeks (=1 cycle) until disease progression or unacceptable toxicities.
  ABTL0812 will be administered daily at its RP2D. ABTL0812 will be administered as single agent during a run-in period of one week before starting the first cycle of FOLFIRINOX, then daily during chemotherapy cycles. Also, ABTL0812 will be maintained once chemotherapy is discontinued, if ABTL0812 is tolerated and if the patient is in response or stable disease.
  Interventions: Drug: ABTL0812; Drug: Folfirinox
- Arm B) PLACEBO + FOLFIRINOX (Experimental): FOLFIRINOX will be dosed according to the standard following regimen:
  * oxaliplatin 85 mg/m2, administered as 2-hour iv infusion
  * leucovorin 400 mg/m2, administered as 2-hour iv infusion
  * irinotecan 180 mg/m2, administered as 1.5-hour iv infusion
  * fluorouracil 2400 mg/m2, administered as 46-hour iv infusion every 2 weeks (=1 cycle) until disease progression or unacceptable toxicities.
  Placebo will be administered at the same volume than ABTL0812 in arm A) FOLFIRINOX, then daily during chemotherapy cycles. Also, placebo will be maintained once chemotherapy is discontinued.
  Interventions: Drug: ABTL0812; Drug: Placebo

INTERVENTIONS:
Drug: ABTL0812 — ABTL0812 will be administered daily at its RP2D. ABTL0812 will be administered as single agent during a run-in period of one week before starting the first cycle of FOLFIRINOX, then daily during chemotherapy cycles. Also, ABTL0812 will be maintained once chemotherapy is discontinued, if ABTL0812 is tolerated and if the patient is in response or stable disease.
Drug: Folfirinox — FOLFIRINOX will be dosed according to the standard following regimen:
  * oxaliplatin 85 mg/m2, administered as 2-hour iv infusion
  * leucovorin 400 mg/m2, administered as 2-hour iv infusion
  * irinotecan 180 mg/m2, administered as 1.5-hour iv infusion
  * fluorouracil 2400 mg/m2, administered as 46-hour iv infusionevery 2 weeks (=1 cycle) until disease progression or unacceptable toxicities.
  Other Names: Chemotherapy
  Arms: Arm A) ABTL0812 + FOLFIRINOX
Drug: Placebo — Placebo will be administered daily at the same regim as ABTL0812. Placebo will be administered as single agent during a run-in period of one week before starting the first cycle of FOLFIRINOX, then daily during chemotherapy cycles. Also, placebo will be maintained once chemotherapy is discontinued, if the patient is in response or stable disease.
  Arms: Arm B) PLACEBO + FOLFIRINOX

SUMMARY:
A Phase I open label followed by a Phase II randomized, controlled study to assess the efficacy and safety of ABTL0812 in combination with FOLFIRINOX for first-line treatment of metastatic pancreatic. Funded by: FDA OOPD (Grant #FD-R-006817-01), H2020 EIC Accelerator (Grant #954825) and Ability Pharmaceuticals SL.

DETAILED DESCRIPTION:
Phase I: This is an open label Phase I to determine the RP2D of ABTL0812 in combination with FOLFIRINOX. All patients will receive ABTL0812 in combination with FOLFIRINOX.

A dose de-escalation phase will be performed in which up to 3 different ABTL0812 dose levels will be tested in combination with FOLFIRINOX. ABTL0812 doses are: 1300 mg tid (starting dose), followed (if necessary) by 975 mg tid and 650 mg tid. Patient intra-escalation is not allowed.

Phase II: This is a double blind, randomized, placebo-controlled Phase II multicenter study to evaluate ABTL0812 in combination with FOLFIRINOX for first-line treatment of metastatic pancreatic cancer. Patients will be randomized to one of two groups: arm A) receiving ABTL0812 in addition to FOLFIRINOX and arm B) receiving FOLFIRINOX plus placebo.

Arm A) ABTL0812 + FOLFIRINOX Arm B) PLACEBO + FOLFIRINOX

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed carcinoma, adenocarcinoma or ductal adenocarcinoma of the pancreas.
2. Confirmed metastatic disease
3. Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 guidelines with at least one "target lesion" to be used to assess response. Tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1.
5. Age, older than 18 years old
6. Adequate hematologic function, measured as:

   * absolute neutrophil count ≥ 1.5x109/L
   * platelet count ≥ 100x109/L without transfusion support
   * hemoglobin ≥ 10 g/dL
7. Total bilirubin ≤ 1.5 x ULN
8. Albumin ≥ 3.3 g/dL
9. AST (SGOT) and ALT (SGPT) ≤ 2.5 times x upper limit of normal (≤ 5 times the ULN in patients with evidence of liver metastases)
10. Alkaline phosphatase ≤ 2.5 times ULN (≤5 times the ULN in patients with evidence of liver metastases)
11. Glomerular filtration rate (GFR) ≥ 60 mL/min/1.73 m2
12. Only for Phase II patients. If available, a sample of tumor tissue or cytology (either archival or new tumor biopsy) for biomarker analyses. The most recently collected tumor tissue sample should be provided.
13. Contraception: All premenopausal female patients must use contraception. Male patients and their female partners (if fertile), must use contraception as well. In both cases, contraception means two forms of highly effective contraception during the study and for a period of 6 months following the last administration of the study drug.
14. Willing and able to provide informed consent
15. Ability and willingness to comply with study visits, treatment, testing, and to comply with the protocol.

Exclusion criteria

1. Patients with any histology other than carcinoma, adenocarcinoma or ductal adenocarcinoma (such as squamous cell, acinar cell, medullary, colloid, neuroendocrine, etc)
2. Patients has only locally advanced disease, resectable or borderline resectable.
3. The patient has received chemotherapy as adjuvant therapy for locally advanced disease, resectable or borderline resectable.
4. Patient has received previous abdominal radiotherapy, (with the exception of analgesic radiotherapy that was not performed on target lesions).
5. Patients previously treated with an inhibitor of the PI3K/Akt/mTOR pathway by a systemic route.
6. History of chronic diarrhea or inflammatory disease of the colon or rectum, or occlusion or sub-occlusion not resolved under symptomatic treatment
7. Patient is pregnant or in lactation period. High sensitivity pregnancy test (urine or serum) to be performed within 7 days before study treatment starts.
8. Patient had myocardial infarction within ≤ 6 months prior to study entry, LVEF <50%, symptomatic congestive heart failure (New York Heart Association > class II), unstable angina pectoris, or unstable cardiac arrhythmia requiring medication.
9. 12-lead ECG with clinically relevant abnormality or showing a QTcF >450 ms, PR >210 ms, or QRS >120 ms at screening.
10. Patients with any other medical conditions (such as psychiatric illness, cardiovascular disease, infectious diseases, abnormal physical examination or laboratory findings) that in the opinion of the investigator may interfere with the planned treatment, affect patient compliance or place the patient at high risk from treatment-related complications.
11. Patient has active Hepatitis B or C, human immunodeficiency virus (HIV) or Covid-19 infection with non-controlled disease according to the treating physician.
12. Patients unable to provide informed consent like those under administrative or legal supervision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Phase I - RP2D | 5 weeks
  Recommended Phase II Dose (RP2D) of ABTL0812 in combination with FOLFIRINOX
Phase II - PFS | 1 year
  PFS using RECIST v1.1 by central review

SECONDARY OUTCOMES:
PFS | 1 year
  PFS using RECIST v1.1 by investigator analysis
ORR | 1 year
  Objective response rate
PFS 6 m | 6 months
  PFS
TTR | 1 year
  Time to response
DOR | 1 year
  Duration of response
OS | 5 years
  Overall survival
OS 1y | 1 year
  Overall survival
Adverse events | 1 year
  Number of participants with Adverse Events (AE). AEs classified according to CTCAE v5.0

OTHER OUTCOMES:
PK - Cmax | 1 month
  Determination of peak plasma concentration
PK - AUC | 1 month
  Determinatoin of Area under the plasma concentration versus time curve
Quality of Life Questionnaire QLC-C30 | 1 year
  Quality of life measured with questionnaires QLC-C30
Quality of Life Questionnaire QLQ-PAN26 | 1 year
  Quality of life measured with questionnaires QLQ-PAN26

CONTACTS AND LOCATIONS:
Overall Officials: Marc Cortal, Study Director — Ability Pharmaceuticals SL
Locations (24):
- United States (4):
  - Cedars Sinai, Los Angeles, California
  - University of Kansas Cancer Center, Westwood, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Cincinnati, Cincinnati, Ohio
- France (3):
  - CGFL Dijon, Dijon
  - Institute Paoli-Calmettes, Marseille
  - Institut Gustave Roussy, Villejuif
- Israel (3):
  - Rabam MC, Haifa
  - Shaare Zedek MC, Jerusalem
  - Sheba MC, Ramat Gan
- Spain (14):
  - ICO Badalona, Badalona, Barcelona
  - Centro Oncológico de Galicia, A Coruña, Galicia
  - Hospital General Universitario Dr. Balmis, Alicante
  - Hospital Quiron Salud, Barcelona
  - Vall d'Hebron University Hospital, Barcelona
  - ICO Girona, Girona
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital Gregorio Marañón, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital General Universitario Morales Meseguer, Murcia
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario de Toledo, Toledo
  - Hospital Universitario de Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Erazo T, Lorente M, Lopez-Plana A, Munoz-Guardiola P, Fernandez-Nogueira P, Garcia-Martinez JA, Bragado P, Fuster G, Salazar M, Espadaler J, Hernandez-Losa J, Bayascas JR, Cortal M, Vidal L, Gascon P, Gomez-Ferreria M, Alfon J, Velasco G, Domenech C, Lizcano JM. The New Antitumor Drug ABTL0812 Inhibits the Akt/mTORC1 Axis by Upregulating Tribbles-3 Pseudokinase. Clin Cancer Res. 2016 May 15;22(10):2508-19. doi: 10.1158/1078-0432.CCR-15-1808. Epub 2015 Dec 15. PMID 26671995
- [Background] Munoz-Guardiola P, Casas J, Megias-Roda E, Sole S, Perez-Montoyo H, Yeste-Velasco M, Erazo T, Dieguez-Martinez N, Espinosa-Gil S, Munoz-Pinedo C, Yoldi G, Abad JL, Segura MF, Moran T, Romeo M, Bosch-Barrera J, Oaknin A, Alfon J, Domenech C, Fabrias G, Velasco G, Lizcano JM. The anti-cancer drug ABTL0812 induces ER stress-mediated cytotoxic autophagy by increasing dihydroceramide levels in cancer cells. Autophagy. 2021 Jun;17(6):1349-1366. doi: 10.1080/15548627.2020.1761651. Epub 2020 May 25. PMID 32397857
- [Background] Felip I, Moiola CP, Megino-Luque C, Lopez-Gil C, Cabrera S, Sole-Sanchez S, Munoz-Guardiola P, Megias-Roda E, Perez-Montoyo H, Alfon J, Yeste-Velasco M, Santacana M, Dolcet X, Reques A, Oaknin A, Rodriguez-Freixinos V, Lizcano JM, Domenech C, Gil-Moreno A, Matias-Guiu X, Colas E, Eritja N. Therapeutic potential of the new TRIB3-mediated cell autophagy anticancer drug ABTL0812 in endometrial cancer. Gynecol Oncol. 2019 May;153(2):425-435. doi: 10.1016/j.ygyno.2019.03.002. Epub 2019 Mar 7. PMID 30853360
- [Background] Lopez-Plana A, Fernandez-Nogueira P, Munoz-Guardiola P, Sole-Sanchez S, Megias-Roda E, Perez-Montoyo H, Jauregui P, Yeste-Velasco M, Gomez-Ferreria M, Erazo T, Ametller E, Recalde-Percaz L, Moragas-Garcia N, Noguera-Castells A, Mancino M, Moran T, Nadal E, Alfon J, Domenech C, Gascon P, Lizcano JM, Fuster G, Bragado P. The novel proautophagy anticancer drug ABTL0812 potentiates chemotherapy in adenocarcinoma and squamous nonsmall cell lung cancer. Int J Cancer. 2020 Aug 15;147(4):1163-1179. doi: 10.1002/ijc.32865. Epub 2020 Feb 6. PMID 31943158
- [Background] Vidal L, Victoria I, Gaba L, Martin MG, Brunet M, Colom H, Cortal M, Gomez-Ferreria M, Yeste-Velasco M, Perez A, Rodon J, Sohal DPS, Lizcano JM, Domenech C, Alfon J, Gascon P. A first-in-human phase I/Ib dose-escalation clinical trial of the autophagy inducer ABTL0812 in patients with advanced solid tumours. Eur J Cancer. 2021 Mar;146:87-94. doi: 10.1016/j.ejca.2020.12.019. Epub 2021 Feb 12. PMID 33588149
- [Background] Paris-Coderch L, Soriano A, Jimenez C, Erazo T, Munoz-Guardiola P, Masanas M, Antonelli R, Boloix A, Alfon J, Perez-Montoyo H, Yeste-Velasco M, Domenech C, Roma J, Sanchez de Toledo J, Moreno L, Lizcano JM, Gallego S, Segura MF. The antitumour drug ABTL0812 impairs neuroblastoma growth through endoplasmic reticulum stress-mediated autophagy and apoptosis. Cell Death Dis. 2020 Sep 17;11(9):773. doi: 10.1038/s41419-020-02986-w. PMID 32943619
- [Background] Mancini A, Colapietro A, Cristiano L, Rossetti A, Mattei V, Gravina GL, Perez-Montoyo H, Yeste-Velasco M, Alfon J, Domenech C, Festuccia C. Anticancer effects of ABTL0812, a clinical stage drug inducer of autophagy-mediated cancer cell death, in glioblastoma models. Front Oncol. 2022 Nov 2;12:943064. doi: 10.3389/fonc.2022.943064. eCollection 2022. PMID 36408162
- [Derived] Polonio-Alcala E, Sole-Sanchez S, Munoz-Guardiola P, Megias-Roda E, Perez-Montoyo H, Yeste-Velasco M, Alfon J, Lizcano JM, Domenech C, Ruiz-Martinez S, Puig T. ABTL0812 enhances antitumor effect of paclitaxel and reverts chemoresistance in triple-negative breast cancer models. Cancer Commun (Lond). 2022 Jun;42(6):567-571. doi: 10.1002/cac2.12282. Epub 2022 Mar 16. No abstract available. PMID 35293148